CLINICAL TRIAL: NCT04743895
Title: Randomized, Single Blinded Pilot Study of Stainless Steel Wire Cerclage Versus FiberTape® Cerclage
Brief Title: Study Comparing Steel Wire to a Flat, Braided Suture to Close the Breastbone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: US-19092
Record Dates: First submitted 2021-02-02; First posted 2021-02-08 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Sternotomy

STUDY DESIGN:
Intervention Model Description: Randomized, Single Blinded Study
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant is blinded to study treatment and radiographers that assess CT scans are also blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Stainless Steel Wire Cerclage (Active Comparator): Sternotomy closure using Stainless Steel Wire Cerclage
  Interventions: Device: Stainless Steel Wire Cerclage
- FiberTape Cerclage (Active Comparator): Sternotomy closure using FiberTape
  Interventions: Device: Stainless Steel Wire Cerclage

INTERVENTIONS:
Device: Stainless Steel Wire Cerclage — Wire cerclage used to close sternum after cardiothoracic surgery.

SUMMARY:
This pilot study is prospective, randomized, single-blinded, single-center for adult patients undergoing sternotomy closure after cardiac surgery. The clinical, patient-reported, and imaging outcomes will be measured comparing standard stainless steel wire (SSW) cerclage versus the FiberTape cerclage.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the progression of sternal healing in subjects that underwent midline sternal closure with FiberTape cerclage compared to subjects that underwent midline sternal closure with stainless steel wire.

The secondary objectives are to evaluate the complication rate and postoperative pain of subjects that underwent midline sternal closure with FiberTape cerclage compared to subjects that underwent midline sternal closure with stainless steel wire.

CT scans are performed at three months postoperatively to assess sternal healing. Two radiologists will read all CT scans. Axial slices are analyzed at five locations along the sternum (manubrium, top of the aortic arch, aortopulmonary window, main pulmonary arteries, and aortic root) using a 6-point quantitative scale (0=no sign of healing, 1=minimal healing, 2=mild healing, 3=moderate healing, 4=partial synthesis, 5=complete synthesis).

All adverse events related to the sternal closure procedure or the devices used for closure will be collected.

Postoperative pain scores will be collected using a 10 cm visual analog scale (VAS) with a numeric rating of 0 to 10. Sternal pain will be rated at rest, coughing, and with movement. Postoperative analgesic use for sternal closure pain will be evaluated.The Veterans Rand (VR-12) health survey will be collected postoperatively (see schedule of events for details).

ELIGIBILITY:
Inclusion Criteria:

1. The subject is age 18 or over.
2. The subject has a planned full median sternotomy.
3. The subject has the ability to read, understand and sign the written informed consent document and complete the online surveys.

Exclusion Criteria:

1. The subject is having a re-operative sternotomy.
2. The subject is having an emergency or salvage operation.
3. The subject has an unplanned sternotomy incision.
4. The subject had an incomplete sternotomy.
5. The subject has chronic pain syndromes or chronic narcotic administration.
6. The subject has a history of chest irradiation.
7. The subject is unwilling to comply with study follow-up visits and surveys.
8. The subject has a sternal infection or suspected sternal infection.
9. The subject has any known comorbidity that will influence the outcomes.
10. The subject is considered vulnerable (i.e. prisoner, child, pregnant, handicapped, or mentally disabled person).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Progression of sternal healing | 3 months post-operative
  A CT scan will be used to assess sternal healing. Axial slices will be analyzed at 5 locations along the sternum using a 6 point quantitative scale. (0-no healing, 1- minimal healing, 2-mild healing, 3-moderate healing, 4-partial synthesis, 5-complete synthesis).

SECONDARY OUTCOMES:
Complication rate | Collected at Immediate post-operatively, again at 3 weeks, 6 weeks, 3 months, 6 months
  Device related adverse event collection
Visual Analog Scale (VAS) | Immediate post-operatively, 3 weeks, 6 weeks, 3 months, 6 months
  Patient reported pain scale using a 10 cm scale with a numeric rating of 0 to 10, with 0 being no pain to 10 being worst pain.
Veteran's Rand Health Survey | Immediate post-operatively, 3 weeks, 6 weeks, 3 months, 6 months
  Patient reported physical and mental health survey. Answers are summarized into 2 scores, a physical component score (PCS) and a mental component score (MCS). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS and MCS are both 50 points. The United States population standard deviation is 10 points. Therefore, each increment of 10 points above or below 50 corresponds to one standard deviation away from the population average.
Analgesic medication Log | Collected at immediate post-operatively during hospital stay, again at 3 weeks, 6 weeks, 3 months and 6 months.
  Analgesic use for sternal pain will be collected on a medication log, tracking type of pain medication, dose and start and ends dates.

CONTACTS AND LOCATIONS:
Locations (1):
- Lee Memorial Health System, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: No